CLINICAL TRIAL: NCT01506115
Title: Observational Study for Safety and Efficacy of Photodynamic Therapy for Bile Duct Invasion of Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Photodynamic Therapy for Bile Duct Invasion of Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-048
Record Dates: First submitted 2011-12-29; First posted 2012-01-09 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2012-01

CONDITIONS: Hepatocellular Carcinoma; Obstructive Jaundice
Keywords: Hepatocellular carcinoma; Obstructive jaundice; Photodynamic therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Jaundice, Obstructive | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HCC with bile duct invasion (Experimental): Photodynamic therapy with biliary drainage in patients with bile duct invasion of unresectable HCC
  Interventions: Drug: Photofrin

INTERVENTIONS:
Drug: Photofrin — Photodynamic therapy: Intravenous Photofrin at a dose of 2 mg/kg body weight, 48 hours before photoactivation by intraluminal light illumination
  Other Names: Photofrin (Axcan Pharma Inc., Mount-Saint-Hilaire, Canada)

SUMMARY:
The prognosis of patients with obstructive jaundice caused by hepatocellular carcinoma (HCC) is dismal even after biliary drainage; due to malfunction of the biliary drainage tube caused by hemobilia and/or tumor emboli. Photodynamic therapy (PDT) in hilar cholangiocarcinoma improves biliary drainage and prolongs survival. The aims of this study were to assess the safety and efficacy of PDT in unresectable HCC with bile duct invasion.

DETAILED DESCRIPTION:
As more therapies are available for patients with hepatocellular carcinoma (HCC), the survival rate has improved. The incidence of jaundice in patients with HCC is reported as 5-44%, and substantial number of patients experience obstructive jaundice. With the improvement of survival in patients with HCC, it is not uncommon to encounter HCC patients with obstructive jaundice in clinical practice.

The prognosis of patients with obstructive jaundice caused by HCC is dismal due to progressive liver failure, rapid tumor progression and ineffective biliary drainage. The mean survival of HCC with obstructive jaundice after biliary drainage ranges from 2.5 to 4.5 months. Effective biliary drainage to improve jaundice and liver function is inevitably needed for further treatment. However, it is difficult to maintain the patency of the bile duct because recurrent obstruction frequently develops due to hemobilia.

Photodynamic therapy (PDT) with biliary drainage is a promising treatment option for advanced cholangiocarcinoma. Presence of the photosensitizer only itself is nontoxic, but showing light with specific wavelengths can induce cytotoxicity. The systemically administrated photosensitizer accumulates preferentially in proliferating tissue. If this targeted lesion is then illuminated by light of a specific wavelength, the activated photosensitizer generates reactive oxygen species, which trigger cell death by apoptosis and necrosis of the cells in the specific area. Experience with PDT in cholangiocarcinoma suggests that a survival benefit can be achieved by prolonged relief of the obstruction.

The investigators hypothesized that conducting PDT with biliary stenting in patients with obstructive jaundice caused by bile duct invasion of HCC would improves stent patency and other clinical outcomes. The aim of this study was to evaluate the safety and efficacy of PDT in HCC patients with bile duct invasion.

ELIGIBILITY:
Inclusion Criteria:

* Known HCC: Diagnosis of HCC based on the 2005 AASLD (American Association for the Study of Liver Diseases) practice guidelines
* Unresectable HCC: Determined based on the BCLC (Barcelona-Clinic-Liver-Cancer) staging and treatment system
* Bile duct invasion of HCC: Confirmed by pathology via endoscopic retrograde cholangiopancreatogram (ERCP) or percutaneous transhepatic biliary drainage (PTBD). In case pathological diagnosis is clinically impossible, confirmed by dynamic CT or MRI showing that typical arterial enhancing mass in dilated bile duct and previous HCC diagnosis.

Exclusion Criteria:

* Severe renal disease
* Severe cardiac disease
* Bleeding tendency
* Porphyria

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Complications associated with the procedure | Six months
  * Procedure related cholangitis: fever accompanied by biliary pain that developed within three days after PDT without other infection
  * Procedure related pancreatitis: abdominal pain and increases in amylase and lipase levels threefold higher than normal
  * Procedure related bleeding: more than a 5% decrease in hematocrit compared to the initial value and coexisting bleeding on abdominal CT or endoscopy
  * Complications associated with the photosensitizer: classified as photosensitivity, burn, and pigmentation

SECONDARY OUTCOMES:
Improvement of jaundice | Six months
  The improvement of jaundice was defined as a decrease in total bilirubin by more than 30% of the pre-procedural value.
Disappearance of hemobilia | Six months
  Disappearance of hemobilia was defined when there was no more evidence of bleeding in patients with previous hemobilia after PDT.
Survival time | Six months
  Survival time was defined as the duration from the date of imaging showing bile duct invasion of HCC to the date of death or to the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Hyuck Lee, M.D., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center 81 Irwon-Ro Gangnamgu, Seoul, South Korea

REFERENCES:
- [Background] El-Serag HB. Hepatocellular carcinoma. N Engl J Med. 2011 Sep 22;365(12):1118-27. doi: 10.1056/NEJMra1001683. No abstract available. PMID 21992124
- [Background] Singal AG, Marrero JA. Recent advances in the treatment of hepatocellular carcinoma. Curr Opin Gastroenterol. 2010 May;26(3):189-95. doi: 10.1097/MOG.0b013e3283383ca5. PMID 20224395
- [Background] Lai EC, Lau WY. Hepatocellular carcinoma presenting with obstructive jaundice. ANZ J Surg. 2006 Jul;76(7):631-6. doi: 10.1111/j.1445-2197.2006.03794.x. PMID 16813631
- [Background] Qin LX, Tang ZY. Hepatocellular carcinoma with obstructive jaundice: diagnosis, treatment and prognosis. World J Gastroenterol. 2003 Mar;9(3):385-91. doi: 10.3748/wjg.v9.i3.385. PMID 12632482
- [Background] Lau WY, Leow CK, Leung KL, Leung TW, Chan M, Yu SC. Cholangiographic features in the diagnosis and management of obstructive icteric type hepatocellular carcinoma. HPB Surg. 2000;11(5):299-306. doi: 10.1155/2000/79241. PMID 10674744
- [Background] Lau WY, Leung JW, Li AK. Management of hepatocellular carcinoma presenting as obstructive jaundice. Am J Surg. 1990 Sep;160(3):280-2. doi: 10.1016/s0002-9610(06)80023-1. PMID 2168129
- [Background] Lau W, Leung K, Leung TW, Liew CT, Chan MS, Yu SC, Li AK. A logical approach to hepatocellular carcinoma presenting with jaundice. Ann Surg. 1997 Mar;225(3):281-5. doi: 10.1097/00000658-199703000-00007. PMID 9060584
- [Background] Cho HC, Lee JK, Lee KH, Lee KT, Paik S, Choo SW, Do YS, Choo IW. Are endoscopic or percutaneous biliary drainage effective for obstructive jaundice caused by hepatocellular carcinoma? Eur J Gastroenterol Hepatol. 2011 Mar;23(3):224-31. doi: 10.1097/MEG.0b013e3283436ff6. PMID 21228705
- [Background] Matsueda K, Yamamoto H, Umeoka F, Ueki T, Matsumura T, Tezen T, Doi I. Effectiveness of endoscopic biliary drainage for unresectable hepatocellular carcinoma associated with obstructive jaundice. J Gastroenterol. 2001 Mar;36(3):173-80. doi: 10.1007/s005350170125. PMID 11291880
- [Background] Chen MF, Jan YY, Jeng LB, Hwang TL, Wang CS, Chen SC. Obstructive jaundice secondary to ruptured hepatocellular carcinoma into the common bile duct. Surgical experiences of 20 cases. Cancer. 1994 Mar 1;73(5):1335-40. doi: 10.1002/1097-0142(19940301)73:53.0.co;2-m. PMID 8111698
- [Background] Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire. A comparison of lipiodol chemoembolization and conservative treatment for unresectable hepatocellular carcinoma. N Engl J Med. 1995 May 11;332(19):1256-61. doi: 10.1056/NEJM199505113321903. PMID 7708069
- [Background] Shim CS, Cheon YK, Cha SW, Bhandari S, Moon JH, Cho YD, Kim YS, Lee LS, Lee MS, Kim BS. Prospective study of the effectiveness of percutaneous transhepatic photodynamic therapy for advanced bile duct cancer and the role of intraductal ultrasonography in response assessment. Endoscopy. 2005 May;37(5):425-33. doi: 10.1055/s-2005-861294. PMID 15844020
- [Background] Zoepf T, Jakobs R, Arnold JC, Apel D, Riemann JF. Palliation of nonresectable bile duct cancer: improved survival after photodynamic therapy. Am J Gastroenterol. 2005 Nov;100(11):2426-30. doi: 10.1111/j.1572-0241.2005.00318.x. PMID 16279895
- [Background] Harewood GC, Baron TH, Rumalla A, Wang KK, Gores GJ, Stadheim LM, de Groen PC. Pilot study to assess patient outcomes following endoscopic application of photodynamic therapy for advanced cholangiocarcinoma. J Gastroenterol Hepatol. 2005 Mar;20(3):415-20. doi: 10.1111/j.1440-1746.2005.03582.x. PMID 15740486
- [Background] Dumoulin FL, Gerhardt T, Fuchs S, Scheurlen C, Neubrand M, Layer G, Sauerbruch T. Phase II study of photodynamic therapy and metal stent as palliative treatment for nonresectable hilar cholangiocarcinoma. Gastrointest Endosc. 2003 Jun;57(7):860-7. doi: 10.1016/s0016-5107(03)70021-2. PMID 12776033
- [Background] Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mossner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology. 2003 Nov;125(5):1355-63. doi: 10.1016/j.gastro.2003.07.015. PMID 14598251
- [Background] Rumalla A, Baron TH, Wang KK, Gores GJ, Stadheim LM, de Groen PC. Endoscopic application of photodynamic therapy for cholangiocarcinoma. Gastrointest Endosc. 2001 Apr;53(4):500-4. doi: 10.1067/mge.2001.113386. PMID 11275896
- [Background] Ortner MA. Photodynamic therapy for cholangiocarcinoma: overview and new developments. Curr Opin Gastroenterol. 2009 Sep;25(5):472-6. doi: 10.1097/MOG.0b013e32832e6e1f. PMID 19550314
- [Background] Kahaleh M, Mishra R, Shami VM, Northup PG, Berg CL, Bashlor P, Jones P, Ellen K, Weiss GR, Brenin CM, Kurth BE, Rich TA, Adams RB, Yeaton P. Unresectable cholangiocarcinoma: comparison of survival in biliary stenting alone versus stenting with photodynamic therapy. Clin Gastroenterol Hepatol. 2008 Mar;6(3):290-7. doi: 10.1016/j.cgh.2007.12.004. Epub 2008 Feb 6. PMID 18255347
- [Background] Witzigmann H, Berr F, Ringel U, Caca K, Uhlmann D, Schoppmeyer K, Tannapfel A, Wittekind C, Mossner J, Hauss J, Wiedmann M. Surgical and palliative management and outcome in 184 patients with hilar cholangiocarcinoma: palliative photodynamic therapy plus stenting is comparable to r1/r2 resection. Ann Surg. 2006 Aug;244(2):230-9. doi: 10.1097/01.sla.0000217639.10331.47. PMID 16858185
- [Background] Hu J, Pi Z, Yu MY, Li Y, Xiong S. Obstructive jaundice caused by tumor emboli from hepatocellular carcinoma. Am Surg. 1999 May;65(5):406-10. PMID 10231205
- [Background] Ikenaga N, Chijiiwa K, Otani K, Ohuchida J, Uchiyama S, Kondo K. Clinicopathologic characteristics of hepatocellular carcinoma with bile duct invasion. J Gastrointest Surg. 2009 Mar;13(3):492-7. doi: 10.1007/s11605-008-0751-0. Epub 2008 Nov 15. PMID 19011945
- [Background] Kubota Y, Seki T, Kunieda K, Nakahashi Y, Tani K, Nakatani S, Yamaguchi T, Mizuno T, Inoue K. Biliary endoprosthesis in bile duct obstruction secondary to hepatocellular carcinoma. Abdom Imaging. 1993;18(1):70-5. doi: 10.1007/BF00201706. PMID 8381692